CLINICAL TRIAL: NCT01517087
Title: Structural and Functional Brain Imaging Markers of Upper Motor Neuron Function
Brief Title: Studying Motor Neuron Tests
Status: Completed | Type: Observational
Sponsor: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 120060; 12-N-0060
Record Dates: First submitted 2012-01-24; First posted 2012-01-25 (Estimated); Last update posted 2021-03-12 (Actual); Status verified 2020-12

CONDITIONS: Healthy Subjects; Magnetic Resonance Imaging; Central Nervous System; Volunteer; Neurological Disorder
Keywords: Cerebrospinal Fluid; Magnetic Resonance Spectroscopy; Transcranial Magnetic Stimulation (TMS); Diffusion Tensor Imaging; Functional Magnetic Resonance Imaging (fMRI); Healthy Volunteer; HV
MeSH Terms: conditions — Nervous System Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- 1: neurologically normal, healthy adults, age 35 or older.

SUMMARY:
Background:

- People with motor neuron disorders have changes in the parts of the brain that control movement. Some tests that are currently used to study these changes are magnetic resonance imaging (MRI) and transcranial magnetic stimulation (TMS). We don t know if MRI scans and TMS give the same results if done at different times in the same person. Researchers want to see if these tests produce different results if given to healthy adults on two separate occasions.

Objectives:

- To test the reliability of different tests of the brain used to study motor neuron disorders.

Eligibility:

* <TAB>Healthy individuals at least 35 years of age who have no history of neurological disorders and take no medications.
* <TAB>Pregnant women may not participate.

Design:

* Participants will be screened with a medical history and physical exam.
* Participants will have two testing visits 1 to 6 months apart.
* The first visit will have three parts. The first part is a neurological exam to test strength, sensation, reflexes, and coordination of movement. The second part will be TMS tests. The third part will involve an MRI scan to study the parts of the brain that control movement.
* At the second visit, participants will have MRI scanning only.

DETAILED DESCRIPTION:
Objective

The objective of the protocol is to determine the test-retest reliability of imaging techniques that measure the structural and functional integrity of the motor cortex in healthy subjects. Our goal is to determine whether such measures are sufficiently reproducible that they may be used to follow disease progression over time in patients with motor neuron disease. A second objective is to obtain age-matched normative data to provide reference values for studies examining the correlation of physiological and clinical measurements of motor function, cognitive testing, and plasma and spinal fluid biomarker measures with disease progression in patients with motor neuron disease.

Study Population

55 neurologically normal, healthy adults, age 35 or older

Design

Each subject will undergo several sessions of testing. The first testing session will consist of a clinical examination with measurements of movement speed. Subjects will undergo one session with transcranial magnetic stimulation of the brain, one session of cognitive testing, and three sessions of magnetic resonance imaging of the brain, one to eighteen months apart. Subjects may opt-in for collection of blood and spinal fluid to provide controls for biomarker studies in motor neuron disease patients.

Outcome Measures

The primary outcome is the test-retest reliability of magnetic resonance imaging measurements of the motor cortex in individual subjects.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Healthy adults aged 35 and older
* No history of a neurological disorder
* Able to give informed consent

EXCLUSION CRITERIA:

* Treatment within the preceding week with medications that affect neuronal excitability, such as antidepressants, sedatives, and drugs for epilepsy or migraine.
* Change in blood pressure medications within the preceding week.
* Metal in the body such as pacemakers, implanted pumps or other implanted electronic devices, some types of dental implants, aneurysm clips (metal clips on the wall of a large artery), metallic prostheses (including metal pins and rods, heart valves, and cochlear implants), permanent eyeliner or shrapnel fragments.
* Pregnancy. Women of childbearing potential will undergo urine pregnancy testing before MRI scanning.
* Fear of confined spaces.
* Serious medical illness.
* Employees or staff in the investigator's section.

Min Age: 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 55 neurologically normal, healthy adults, age 35 or older.
Sampling Method: Non-Probability Sample
Enrollment: 47 (Actual)
Dates: Start 2012-02-01 (Actual); Primary Completion 2020-11-25 (Actual); Study Completion 2020-11-25 (Actual)

PRIMARY OUTCOMES:
Test-retest reliability of MRI measures | 09/30/2019
  The test-retest reliability will be assessed by calculating the intraclass correlation coefficient (ICC) between the two sessions. An ICC > 0.8 is considered to indicate excellent reliability.

CONTACTS AND LOCATIONS:
Overall Officials: Mary Kay Floeter, M.D., Principal Investigator — National Institute of Neurological Disorders and Stroke (NINDS)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Ellis CM, Simmons A, Jones DK, Bland J, Dawson JM, Horsfield MA, Williams SC, Leigh PN. Diffusion tensor MRI assesses corticospinal tract damage in ALS. Neurology. 1999 Sep 22;53(5):1051-8. doi: 10.1212/wnl.53.5.1051. PMID 10496265
- [Background] Tartaglia MC, Laluz V, Rowe A, Findlater K, Lee DH, Kennedy K, Kramer JH, Strong MJ. Brain atrophy in primary lateral sclerosis. Neurology. 2009 Apr 7;72(14):1236-41. doi: 10.1212/01.wnl.0000345665.75512.f9. PMID 19349603
- [Background] Wong JC, Concha L, Beaulieu C, Johnston W, Allen PS, Kalra S. Spatial profiling of the corticospinal tract in amyotrophic lateral sclerosis using diffusion tensor imaging. J Neuroimaging. 2007 Jul;17(3):234-40. doi: 10.1111/j.1552-6569.2007.00100.x. PMID 17608909
- [Derived] Clark MG, Smallwood Shoukry R, Huang CJ, Danielian LE, Bageac D, Floeter MK. Loss of functional connectivity is an early imaging marker in primary lateral sclerosis. Amyotroph Lateral Scler Frontotemporal Degener. 2018 Nov;19(7-8):562-569. doi: 10.1080/21678421.2018.1517180. Epub 2018 Oct 9. PMID 30299161
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2012-N-0060.html